CLINICAL TRIAL: NCT04113967
Title: Efficacy of a Biodanza Program in People With Alzheimer's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, María del Mar Lopez-Rodriguez, Director, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Universidad de Almería
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer Dementia (AD); Mental Disorder; Mood Disorders; Physically Disabled
Keywords: Biodanza; Alzheimer Dementia; dance therapy; complementary therapies; physical activity
MeSH Terms: conditions — Alzheimer Disease; Mental Disorders; Mood Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodanza Group (Experimental): The biodanza program will consist of 12 sessions, one per week, during three months. Each session will last approximately 60 minutes and an introductory phase (10-15 minutes) and an experience phase (45 minutes) will be divided. It involves moving / dancing according to the suggestions of the monitor and the rhythm of the music.
  Interventions: Other: Biodanza program
- Treatment as usual Group (No Intervention): The control group will continue with its usual treatment and activities, without suffering any alteration. A measurement of the groups (control group and biodanza group) will be carried out before the start and after the end of the sessions.

INTERVENTIONS:
Other: Biodanza program — Biodanza is a form of intervention aimed at promoting health and well-being through the promotion of self-expression and self-regulation through interaction through music and dance. The music accompanied by the movement of the body induces some experiences that present the ability to modify the organism itself both at an organic level, as affective-motor and existential. This intervention constitutes a means for the correct development of human qualities, whose purpose is to integrate the potentials of bond, health and harmony, as well as to develop new alternatives for the life of each individual.
  Other Names: Biodance
  Arms: Biodanza Group

SUMMARY:
This study aims to know the efficacy of a biodanza program in adults diagnosed with Alzheimer's, and it is a randomized controlled trial where the control group, which maintains its usual treatment, will form a waiting list to perform any of the treatments outside the follow-up period. There will also be a group that will carry out intervention with biodanza.

For the selection of the sample, there will be the participation of different Alzheimer associations and geriatric centers in the province of Almeria. The inclusion criteria will be between 60 and 75 years old, with a primary diagnosis of Alzheimer's disease, and who have never participated in any biodanza session or have knowledge about it. Those whose diagnosis is different from Alzheimer's disease or who suffers from a physical or psychological illness that prevents the execution of the sessions and all who do not participate in at least 75% (9 sessions) of the sessions will be excluded from the study.

The biodanza program will consist of 12 sessions, one per week, during three months. The control group will continue with its usual treatment and activities, without suffering any alteration. A measurement of the groups (control group and biodanza group) will be carried out before the start and after the end of the sessions. The questionnaires and scales administered to the participants include demographical and clinical variables, physical state variables, cognitive variables, and emotional and behavioral variables. Finally, statistical analyzes will be performed using SPSS version 23. In the case of quantitative variables, they will be expressed as mean and standard deviation and, when the variables are of qualitative type, they will be represented by frequency and percentages.

DETAILED DESCRIPTION:
Dementia is considered a severely disabling illness for those who suffer from it and is usually devastating for their family and caregivers. It is a syndrome mainly of a chronic or progressive nature, caused by a series of brain diseases that affect memory, behavior, thinking and ability to perform activities of daily living (WHO, 2013).

This study aims to know the efficacy of a biodanza program in adults diagnosed with Alzheimer's.

This is a randomized controlled trial where the control group, which maintains its usual treatment, will form a waiting list to perform any of the treatments outside the follow-up period. There will also be a group that will carry out intervention with biodanza.

In this study, adults with Alzheimer's disease will participate voluntarily, regardless of race or sex. For the selection of the sample, there will be the participation of different Alzheimer associations and geriatric centers in the province of Almeria. The inclusion criteria will be between 60 and 75 years old, with a primary diagnosis of Alzheimer's disease, and who have never participated in any biodanza session or have knowledge about it. Those whose diagnosis is different from Alzheimer's disease or who suffers from a physical or psychological illness that prevents the execution of the sessions and all who do not participate in at least 75% (9 sessions) of the sessions will be excluded from the study.

In accordance with the principles of the Declaration of Helsinki (2013), before the start of the investigation, participants will be informed and sign consent. Subjects will have the right to refuse to participate as well as to withdraw at any time during the study. They will also be assured of complete confidentiality of the data.

The biodanza program will consist of 12 sessions, one per week, during three months. Each session will last approximately 60 minutes and an introductory phase (10-15 minutes) and an experience phase (45 minutes) will be divided. It involves moving / dancing according to the suggestions of the monitor and the rhythm of the music. The control group will continue with its usual treatment and activities, without suffering any alteration. A measurement of the groups (control group and biodanza group) will be carried out before the start and after the end of the sessions. The questionnaires and scales administered to the participants are classified according to the variables to be measured:

DEMOGRAPHICAL AND CLINICAL VARIABLES, including age, sex, family situation, economic level, nationality, employment status, year of diagnosis of the disease, history of the disease and pharmacological treatment. PHYSICAL STATE VARIABLES, including anthropometric measures such as weight, size, and body mass index (BMI) and physical tests through the 6-minute walk test and Tinetti scale. COGNITIVE VARIABLES, through Mini Mental Status Examination (MMSE), Daily Living Activities Index Barthel, and Pfeiffer Short Portable Mental Status Questionnaire. EMOTIONAL AND BEHAVIORAL VARIABLES, using Hamilton Depression Rating Scale, and Pittsburg Sleep Quality Index.

Finally, statistical analyzes will be performed using SPSS version 23. In the case of quantitative variables, they will be expressed as mean and standard deviation and, when the variables are of qualitative type, they will be represented by frequency and percentages.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of Alzheimer's disease,
* never participated in any biodanza session or have knowledge about it.

Exclusion Criteria:

* diagnosis is different from Alzheimer's disease
* suffering from a physical or psychological illness that prevents the execution of the sessions
* do not participate in at least 75% (9 sessions) of the sessions.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 3 months
  The 6MWT is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes. It evaluates the global and integrated responses of all the systems involved during exercise. The self-paced 6MWT assesses the submaximal level of functional capacity. Because most activities of daily living are performed at submaximal levels of exertion, the 6MWD may better reflect the functional exercise level for daily physical activities.
Tinetti test | 3 months
  The Tinetti-test was published by Mary Tinetti (Yale University) to assess the gait and balance in older adults. It is a very good indicator of the fall risk of an individual. The test requires a hard armless chair, a stopwatch and also, a 15feet even and uniform walkway. It has 2 sections; one assesses balance abilities in a chair and also in standing, and the other assesses dynamic balance during gait on a 15feet walkway.The patient is to sit in an armless chair and will be asked to rise up and stay standing. The patient will then turn 360° and then sit back down.This is to test the patients' balance. Next, the patient will have to walk a few meters at a normal speed, followed by turning and walking back at a "fast but safe" speed. The patient will then sit back down. During this test, the patient can use any assistive devices (walking stick, crutches, zimmer frame) they would normally use.
Mini Mental State Examination (MMSE) | 3 months
  The Mini-Mental State Examination (MMSE) is a 10-minute measure of impaired thinking. The summed score of the individual items indicates the current severity of cognitive impairment. Deterioration in cognition is indicated by decreasing scores of repeated tests. The items of the MMSE include tests of orientation, registration, recall, calculation and attention, naming, repetition, comprehension, reading, writing and drawing. Level of consciousness is rated on a scale from coma to fully alert, but the consciousness rating is not summed with the other items. If all items are answered correctly, the score is 30. The mean score for a community-dwelling population over 65 years of age is 27, with a standard deviation of 1.71. Alzheimer's disease patients lose 3-4 points per year of illness after the onset of memory disturbance, although there is wide variability in this phenomenon.
Daily Living Activities Index (Barthel Scale/Index) | 3 months
  The Barthel Scale/Index is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently. The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL (feeding, personal toileting, bathing, dressing and undressing, getting on and off a toilet, controlling bladder, controlling bowel, moving from wheelchair to bed and returning, walking on level surface, or propelling a wheelchair if unable to walk, and ascending and descending stairs). Each item is rated in terms of whether the patient can perform the task independently, with some assistance, or is dependent on help based on observation (0=unable, 1=needs help, 2=independent). The final score is x 5 to get a number on a 100 point score.
Pfeiffer Short Portable Mental Status Questionnaire | 3 months
  Pfeiffer Test is also known as "short portable mental status questionnaire" and abbreviated as "SPMSQ". This questionnaire is an instrument to assess the organic brain deficit, easy to use, reliable, valid and brief, since it consists of 10 questions. The test Pfeiffer assigns a score from 0 to 10, depending on the amount of incorrect questions answered, assigning one point for each incorrect question. Then, on the basis of the errors made, these 10 questions measure the cognitive deterioration and determine its degree through four levels as follows: (0-2 points) normal, (3-4) light, (5-7 points), moderate and (8-10 points) severe.
Hamilton Depression Rating Scale | 3 months
  The Hamilton Rating Scale for Depression, is a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. Although the Hamilton Rating Scale for Depression form lists 21 items, the scoring is based on the first 17. It generally takes 15-20 minutes to complete the interview and score the results. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2.
Pittsburg Sleep Quality Index. | 3 months
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.Traditionally, the items from the PSQI have been summed to create a total score to measure overall sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: No